CLINICAL TRIAL: NCT02476994
Title: A Randomized, Double-Blind, Controlled, Clinical Trial to Evaluate the Risk of Developing Essential Fatty Acid Deficiency in Pediatric Patients, Including Neonates, Receiving Either Clinolipid (Lipid Injectable Emulsion, USP) 20% or Standard-of-Care Soybean Oil-Based Lipid Emulsion
Brief Title: Pediatric Study to Evaluate Risk of Developing Essential Fatty Acid Deficiency When Receiving Clinolipid or Standard-of-Care Lipid Emulsion
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Based on feedback from FDA
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6344-001
Record Dates: First submitted 2015-06-16; First posted 2015-06-22 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Essential Fatty Acid Deficiency (EFAD)
Keywords: Essential Fatty Acids (EFA); Parenteral Nutrition; Clinolipid/Clinoleic; Parenteral Nutrition Associated Cholestasis (PNAC); Parenteral Nutrition Associated Liver Disease (PNALD); Intestinal Failure Associated Liver Disease (IFALD); Phytosterols; Intralipid; Infants/Preterm Infants; FADS1 and FADS2; Short Bowel Syndrome; Cancer Nutrition; Olive Oil Emulsion; Soybean Oil Emulsion
MeSH Terms: conditions — Hyperphagia; Pena Shokeir syndrome, type 1; Short Bowel Syndrome | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinolipid (lipid injectable emulsion, USP) 20% (Experimental): Dosing schedule based on subject's age, weight, and medical condition and as per ESPEN-ESPHAN guidelines.
  Interventions: Drug: Clinolipid
- Intralipid 20% (lipid injectable emulsion, USP) (Active Comparator): Dosing schedule based on subject's age, weight, and medical condition and as per ESPEN-ESPHAN guidelines.
  Interventions: Drug: Intralipid

INTERVENTIONS:
Drug: Clinolipid
  Arms: Clinolipid (lipid injectable emulsion, USP) 20%
Drug: Intralipid — Standard-of-Care Soybean Oil-Based Lipid Emulsion
  Arms: Intralipid 20% (lipid injectable emulsion, USP)

SUMMARY:
This will be a descriptive study designed to evaluate the propensity for hospitalized pediatric patients treated adequately with Clinolipid or standard of care for up to 90 days to develop Essential Fatty Acid Deficiency (EFAD). Additionally, this study design will evaluate the safety and efficacy of using Clinolipid in a pediatric population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients and/or their legal representative must be able to understand the study and voluntarily sign the ICF
2. Patients age <18 years
3. Patients who are able to adhere to protocol requirements
4. Patients who are expected to require PN for at least 7 days
5. Premature infants (<36 weeks of gestation) require at least 80% PN to meet nutrition requirements at study entry; full term infants and children require at least 70% PN to meet nutrition requirements at study entry

Exclusion Criteria:

1. Patients who are not expected to survive hospitalization or with a severe illness with foreseeable intercurrent events that could jeopardize the patient's participation in the study
2. Patients with a known hypersensitivity to lipid emulsion, egg or soybean proteins, or any of the active substances, excipients, or components of the container
3. Patients with a diagnosis of shock, renal failure requiring dialysis, or severe metabolic acidosis (eg, pH <7.10, serum bicarbonate level ≤15 mEq/L , and/or an Anion Gap >16 mEq/L)
4. Patients with hemodynamic instability as judged by the Investigator
5. Patients with uncorrected metabolic disorders (eg, diabetes) or liver disease including cholestasis
6. Patients with severe hyperlipidemia or severe disorders of lipid metabolism characterized by hypertriglyceridemia (triglyceride >400 mg/dL)
7. Patients who are unable to tolerate the necessary laboratory monitoring
8. Patients who have a new and active infection (as assessed by the investigator) at time of initiation of study treatment
9. Patients who are enrolled in another clinical trial involving an investigational agent
10. Patients who were treated with IV lipids within 48 hours of randomization into the study

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baxter Healthcare Corporation, Study Director — Baxter Healthcare Corporation
Locations (4):
- United States (4):
  - Advocate Children's Hospital, Park Ridge, Illinois
  - Riley Hospital for Children at Indiana Health, Indianapolis, Indiana
  - Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Medical University of SC, Neonatology, Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinolipid (Lipid Injectable Emulsion, USP) 20%: Dosing schedule based on subject's age, weight, and medical condition and as per ESPEN-ESPHAN guidelines.
  Clinolipid
Period: Overall Study
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Based on feedback from FDA | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP) | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Essential Fatty Acid Deficiency (EFAD)
Description: Holman Index Calculation
Time Frame: Up to 90 Days
Population: Due to early termination of the study, no formal analysis was conducted.
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Parenteral Nutrition-Associated Cholestasis (PNAC)
Time Frame: Up to 90 Days
Population: Due to early termination of the study, no formal analysis was conducted.
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Genetic Polymorphisms in Fatty Acid Desaturase Genes FADS1 and FADS2
Time Frame: Baseline
Population: Due to early termination of the study, no formal analysis was conducted.
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Fatty Acid Profile
Time Frame: Up to 90 Days
Population: Due to early termination of the study, no formal analysis was conducted.
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Weight
Time Frame: Up to 90 Days
Population: Due to early termination of the study, no formal analysis was conducted.
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phytosterol, Cholesterol, and Squalene Levels
Time Frame: Up to 90 Days
Population: Due to early termination of the study, no formal analysis was conducted.
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline of Hepatic Integrity (ALP, AST, ALT, GGT, Total and Direct Bilirubin)
Time Frame: Up to 90 Days
Population: Due to early termination of the study, no formal analysis was conducted.
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Prescribed and Actual (Total Calories From PN and Oral) Nutritional Intake
Time Frame: Up to 90 Days
Population: Due to early termination of the study, no formal analysis was conducted.
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Vital Signs
Time Frame: Up to 90 Days
Population: Due to early termination of the study, no formal analysis was conducted.
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Adverse Events and Serious Adverse Events
Time Frame: Up to 30 Days After Subject's Last Study Treatment
Population: Due to early termination of the study, no formal analysis was conducted.
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Clinical Laboratory Tests
Time Frame: Up to 90 Days
Population: Due to early termination of the study, no formal analysis was conducted.
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Clinolipid (Lipid Injectable Emulsion, USP) 20% | Intralipid 20% (Lipid Injectable Emulsion, USP)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No